CLINICAL TRIAL: NCT01749462
Title: Oxis 9mcg Turbuhaler Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5127L00001
Record Dates: First submitted 2012-12-12; First posted 2012-12-13 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease,; COPD,; Oxis,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Oxis

SUMMARY:
The purpose of the investigation is to confirm the ADR development and the contributing factors possibly having an impact on the safety under the post-marketing actual use of Oxis 9 mcg Turbuhaler.

DETAILED DESCRIPTION:
Oxis 9mcg Turbuhaler Clinical Experience Investigation

ELIGIBILITY:
Inclusion Criteria:

- Patients treated with Oxis for the first time due to 'relief of various symptoms associated with airway obstructive disorders of chronic obstructive pulmonary disease (Chronic bronchitis, Pulmonary emphysema), which is the indication of this drug.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Oxis for the first time due to 'relief of various symptoms associated with airway obstructive disorders of chronic obstructive pulmonary disease (Chronic bronchitis, Pulmonary emphysema), which is the indication of this drug.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — Astrazeneca KK
Locations (41):
- Japan (41):
  - Research Site, Aichi, D5127l00001
  - Research Site, Akita, D5127l00001
  - Research Site, Aomori, D5127l00001
  - Research Site, Chiba, D5127l00001
  - Research Site, Fukuoka, D5127l00001
  - Research Site, Fukushima, D5127l00001
  - Research Site, Gifu, D5127l00001
  - Research Site, Gunma, D5127l00001
  - Research Site, Hiroshima, D5127l00001
  - Research Site, Hokkaido, D5127l00001
  - Research Site, Hyōgo, D5127l00001
  - Research Site, Ibaraki, D5127l00001
  - Research Site, Ishikawa, D5127l00001
  - Research Site, Kagawa, D5127l00001
  - Research Site, Kagoshima, D5127l00001
  - Research Site, Kanagawa, D5127l00001
  - Research Site, Kochi, D5127l00001
  - Research Site, Kyoto, D5127l00001
  - Research Site, Mie, D5127l00001
  - Research Site, Miyagi, D5127l00001
  - Research Site, Miyazaki, D5127l00001
  - Research Site, Nagano, D5127l00001
  - Research Site, Nagasaki, D5127l00001
  - Research Site, Nara, D5127l00001
  - Research Site, Niigata, D5127l00001
  - Research Site, Numakunai, D5127l00001
  - Research Site, Okayama, D5127l00001
  - Research Site, Okinawa, D5127l00001
  - Research Site, Osaka, D5127l00001
  - Research Site, Ōita, D5127l00001
  - Research Site, Saitama, D5127l00001
  - Research Site, Shiga, D5127l00001
  - Research Site, Shimane, D5127l00001
  - Research Site, Shizuoka, D5127l00001
  - Research Site, Tochigi, D5127l00001
  - Research Site, Tokushima, D5127l00001
  - Research Site, Tokyo, D5127l00001
  - Research Site, Toyama, D5127l00001
  - Research Site, Yamagata, D5127l00001
  - Research Site, Yamaguchi, D5127l00001
  - Research Site, Yamanashi, D5127l00001

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=471&filename=OXS_CSRsynopsis.pdf